CLINICAL TRIAL: NCT06200636
Title: Edge AI-deployed DIGItal Twins for PREDICTing Disease Progression and Need for Early Intervention in Infectious and Cardiovascular Diseases Beyond COVID-19 - Investigation of Biomarkers in Dermal Interstitial Fluid
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Laurenz Kopp Fernandes, Senior physician, Transplant Outpatient Unit, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DIGIPREDICT-Bio
Record Dates: First submitted 2024-01-09; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional group (Experimental): This arm inclcudes all study participants.
  Interventions: Device: Use of the PELSA System for dISF extraction

INTERVENTIONS:
Device: Use of the PELSA System for dISF extraction — Dermal interstitial fluid will be extracted using the investigational device, for further analysis.

SUMMARY:
The study will investigate, if inflammatory and cardio-circulatory biochemical biomarkers are detectable in dermal interstitial fluid (dISF) of heart failure patients, and if there are detectable kinetics of these biomarkers during a cardiopulmonary exercise test. For dISF extraction the PELSA System - an investigational device - will be used.

ELIGIBILITY:
Inclusion Criteria:

* Subject suffers from heart failure (according to ESC 2021 Heart Failure Guidelines).
* Age of subject is ≥18 years.
* Subject is female or male.
* Signed written informed consent.
* For female subjects:

  1. Confirmed post-menopausal state, defined as amenorrhea for at least 12 months, or
  2. If being of childbearing potential:

     1. Negative highly sensitive urine or serum pregnancy test before inclusion, and
     2. Practicing a highly effective birth control method (failure rate of less than 1%):

        1. combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral/intravaginal/ transdermal), or
        2. progestogen-only hormonal contraception associated with inhibition of ovulation (oral/injectable/implantable), or
        3. intrauterine device (IUD), or
        4. intrauterine hormone-releasing system (IUS), or
        5. bilateral tubal occlusion, or
        6. vasectomised partner, or
        7. heterosexual abstinence.
* Subject is capable to perform cardiopulmonary exercise testing.

Exclusion Criteria:

* Subject is breastfeeding.
* Subject suffers from an addiction or from a disease that prevents the subject from recognizing nature, scope, and consequences of the study.
* Subject is treated with immunosuppressive drugs at enrolment.
* Subject requires renal replacement therapy.
* Subject has a known colonisation or infection with multi-drug-resistant pathogens.
* Subject has an open wound in or near the sampling area.
* Subject has any type of tattoo or piercing anywhere in or near the sampling area.
* Subject shows an inability to comply with all the study procedures and follow-up visits.
* Subject is unwilling to consent to saving and propagation of pseudonymised medical data for study reasons.
* Subject is legally detained in an official institution.
* Subject is dependent on the sponsor, the investigator or the study sites.
* Subject participates in a study according to AMG/CTR that investigates immunosuppressive or anticoagulant drugs at the time of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Detection of inflammatory and cardio-circulatory biochemical biomarkers in dermal interstitial fluid of heart failure patients | Before, immediate after and 30 min after a cardiopulmonary exercise test.
  Level above the limit of quantification of the investigated biomarkers in dermal interstitial fluid.

SECONDARY OUTCOMES:
Relationship between the levels of biochemical inflammatory and cardio-circulatory biomarkers in dermal interstitial fluid and their blood levels in heart failure patients. | Before, immediate after and 30 min after a cardiopulmonary exercise test.
  Dermal interstitial fluid levels and blood levels of the investigated biomarkers.
Kinetics of inflammatory and cardio-circulatory biochemical biomarker levels in dermal interstitial fluid and in blood of heart failure patients during exercise testing. | Before, immediate after and 30 min after a cardiopulmonary exercise test.
  Increase or decrease of the levels of the investigated biomarkers in dermal interstitial fluid and in blood during exercise.
Relationship between kinetics of inflammatory and cardio-circulatory biochemical biomarker levels in dermal interstitial fluid and in blood of heart failure patients during exercise testing. | Before, immediate after and 30 min after a cardiopulmonary exercise test.
  Dermal interstitial fluid level change (to first or previous measurement) and blood level change (to first or previous measurement) of the investigated biomarkers during exercise.
Performance of the PELSA system in relation to its intended use. | Before, immediate after and 30 min after a cardiopulmonary exercise test.
  Evidence that the PELSA system can extract interstitial fluid from the skin.
Safety of the PELSA system in relation to its intended use. | Before, immediate after and 30 min after a cardiopulmonary exercise test.
  Documentation of adverse events and serious adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Deutsches Herzzentrum der Charité, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No